CLINICAL TRIAL: NCT05415345
Title: Study on the Immunogenicity and Safety of Co-immunization With Recombinant Human Papillomavirus 16/18 Bivalent Vaccine and Hepatitis E Vaccine
Brief Title: Immunogenicity and Safety of Co-immunization With Cecolin and Hecolin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xiamen Innovax Biotech Co., Ltd (Industry)
Collaborators: Zhejiang Provincial Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROPMHP001
Record Dates: First submitted 2022-05-27; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-05

CONDITIONS: Human Papilloma Virus Infection Type 16; Human Papilloma Virus Infection Type 18; Hepatitis E Virus Infection
MeSH Terms: conditions — Hepatitis E | interventions — hecolin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Participants in this arm will be simultaneously administrated with HPV and HEV vaccine. The immunization schedule is 0,1,6 months.
  Interventions: Biological: Cecolin; Biological: Hecolin
- Group B (Active Comparator): Participants in this arm will be administrated with HPV vaccine. The immunization schedule is 0,1,6 months.
  Interventions: Biological: Cecolin
- Group C (Active Comparator): Participants in this arm will be administrated with HEV vaccine. The immunization schedule is 0,1,6 months.
  Interventions: Biological: Hecolin

INTERVENTIONS:
Biological: Cecolin — Bivalent HPV Vaccine
  Arms: Group A; Group B
Biological: Hecolin — Hepatitis E vaccine
  Arms: Group A; Group C

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of co-immunization with recombinant human papillomavirus bivalent (Types 16,18) vaccine (Escherichia coli) and Hepatitis E vaccine (Escherichia coli)

DETAILED DESCRIPTION:
Cecolin is the first Chinese domestic human papillomavirus (HPV) vaccine. Cecolin is designed to protect against HPV types 16 and 18, the most common virus types that lead to cervical cancer. Hecolin is the first prophylactic vaccine against hepatitis E virus (HEV). The purpose of this study is to evaluate the immunogenicity and safety of co-immunization with Cecolin and Hecolin.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged between 18 and 25 years (including 18 and 25 years) on the day of enrollment
* Judged as healthy and eligible for vaccination by the investigators through a self- reported medical history and some physical examinations
* Willing to participate in this study and sign informed consent form
* Able to understand this study information and willing to comply with all study requirements
* Axillary temperature ≤37.0 °C
* Negative urine pregnancy test

Exclusion Criteria:

* Women who are pregnant or breastfeeding or who plan to get pregnant within the next seven months
* Use of any investigational product or non-registered product (drug or vaccine) within 30 days preceding the first dose of the study vaccine or plan to use during the study period
* Received immunosuppressed, immunoregulation therapy or corticosteroid systemic therapy for more than 14 days in the 6 months before entry, except local treatment
* Administration of any immunoglobulin or blood products within 3 months preceding the first dose of the study vaccine,or plan to use during the study period
* Administration of any inactivated vaccines within 14 days preceding the first dose of the study or attenuated live vaccines within 21 days preceding the first dose of the study
* Had a fever (axillary temperature over 38°C) within 3 days or acute illness requiring systemic antibiotics or antiviral treatment within 5 days before vaccination
* Plan to participate in another clinical study at the same time during the study
* Previous vaccination against HPV or HEV
* Immunodeficiency (such as HIV positive), primary disease of important organs, malignant tumor, .or any immune disease (such as systemic lupus erythematosus, arthritis pauperum, splenectomy or functional asplenia or other disease which might affect immune response)
* History of allergic disease or history of serious adverse events occurring after vaccination, i.e., allergy, urticaria, dyspnea, angioneurotic edema or abdominal pain
* Asthma, which has been unstable for the past two years and requires urgent treatment, hospitalization, oral or intravenous corticosteroid
* Complicated with serious medical diseases, such as hypertension, heart disease, diabetes, hyperthyroidism, etc
* Medical diagnosis of abnormal coagulation function (such as coagulation factor deficiency, coagulation disorders, platelet abnormalities) or coagulation disorders
* Epilepsy, excluding febrile epilepsy under 2 years of age, alcoholic epilepsy 3 years before abstinence or simple epilepsy that did not require treatment for the past 3 years
* Past or present mental illness due to a psychological condition that does not comply with the requirements of the study; mental illness that has not been well controlled in the past two years; mental illness requiring medication; and suicidal tendency in the past five years
* Other medical, psychological, social or occupational factors that, according to the investigators' judgment,might affect the individual's ability to obey the protocol or sign the informed consent.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-06-10 (Estimated)

PRIMARY OUTCOMES:
evaluate the concentration of IgG antibodies to HPV-16 | At 7 months after first dose
  Detect the level of IgG antibodies to HPV-16 at 7 month to determine whether group A is non-inferior to group B
evaluate the concentration of IgG antibodies to HPV-18 | At 7 months after first dose
  Detect the level of IgG antibodies to HPV-18 at 7 month to determine whether group A is non-inferior to group B
evaluate the concentration of IgG antibodies to HEV | At 7 months after first dose
  detect the level of IgG antibodies to HEV at 7 month to determine whether group A is non-inferior to group C

SECONDARY OUTCOMES:
Local and systematic adverse events/reactions occurred within 7 days after each vaccination | During the 7-day period following each vaccination
  Adverse reactions associated with vaccine will be observed in subjects after vaccination. To evaluate number of adverse events/reactions compared with non-simultane vaccination group.
Adverse events/reactions occurred within 30 days after each vaccination | Within 30 days after any vaccination
  To evaluate number of adverse events/reactions compared with non-simultane vaccination group.
Serious adverse events occurred throughout the study | Up to 7 months
  Safety analysis. To evaluate number of SAEs compared with the non-simultane vaccination group

CONTACTS AND LOCATIONS:
Overall Officials: Zhenggang Jiang, Principal Investigator — Zhejiang Provincial Center for Disease Control and Prevention
Locations (1):
- Zhejiang Provincial Center for Disease Control and Prevention, Hanzhou, Zhejiang, China

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263